CLINICAL TRIAL: NCT06076811
Title: Danish Assessment of Minimal Residual Disease by Liquid Biopsies
Brief Title: DANISH.MRD: Danish Assessment of Minimal Residual Disease by Liquid Biopsies
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DANISH.MRD
Record Dates: First submitted 2023-10-04; First posted 2023-10-11 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Neoplasms; Colorectal Cancer; Colorectal Adenocarcinoma; Colorectal Cancer Stage I; Colorectal Cancer Stage II; Colorectal Cancer Stage III
Keywords: Circulating tumor DNA; Surveillance; Risk stratification; Recurrence detection
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue
  Normal tissue
  Whole blood (processed to plasma, buffycoat and serum)
  Dried blood spots.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Approximately two-thirds of all colorectal cancer patients undergo surgery with the aim of curing them. However, despite the surgery, 20-25% of them experience relapse. It is possible to reduce the risk of relapse with chemotherapy, but as chemotherapy is associated with significant side effects, it is only given to patients at high risk of relapse. Currently, the risk is assessed based on an examination of the removed tumor tissue.

In a previous research project, blood samples were taken after patients' surgery and examined for the presence of circulating tumor DNA (ctDNA). When cancer cells in solid tumors die, they release DNA, which can be detected in the blood. DNA in the blood has a half-life of less than 2 hours, so if ctDNA is found in a blood sample taken, e.g., 14 days after surgery, the patient most likely still has cancer cells in their body.

The results show that if a patient has ctDNA in their blood after surgery, the risk of relapse is high. The presence of ctDNA in the blood has the potential to be a better indicator of the risk of future relapse than the tumor examination used today. Therefore, ctDNA analysis has the potential to become a marker that will be used in the future clinical setting for monitoring colorectal cancer.

The overall objective of this study is to confirm that ctDNA found in a blood sample after intended curative treatment for CRC is a marker of residual disease and risk of recurrence and is applicable in clinical practice.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common cancer worldwide. Approximately 75% of patients initially present with potentially curable disease, but despite curatively intended treatment up to 25 % of them experience a relapse of the disease. Upon diagnosis, survival of CRC can be improved by offering adjuvant chemotherapy to patients with a high risk of recurrence, or by early detection of recurrence enabling early intervention which improves patient survival significantly. To achieve this, it is essential to have sensitive and specific tools for correctly identifying patients with a high risk of recurrence and the need for adjuvant therapy, and for early detection of recurrence facilitating early intervention. Non-invasive analysis of circulating tumor DNA (ctDNA) is an emerging tool that has this potential.

Objectives

The overall objective of the study is to confirm that ctDNA detected after intended curative treatment for CRC is a marker of residual disease and risk of recurrence and is applicable in clinical practice.

Primary objectives

P1: To determine the prognostic value of a patient's ctDNA status and compare it with other known prognostic factors. Specifically, the aim is to determine the association between 3-year disease-free survival (DFS) and ctDNA detection status immediately after 1) curative-intended surgery and 2) adjuvant chemotherapy.

P2: To identify a cohort of UICC stage III CRC patients with planned adjuvant chemotherapy. These patients will be offered enrollment in the DANISH.MRD part II (Secondary objective 1 (S1)), and will further be included in a European collaboration named GUIDE.MR-01-CRC, funded by the European Union via the Innovative Health Initiative.

Secondary objectives

S1: To technically assess, compare, and rank commercial ctDNA diagnostics and evaluate their performance after intended-curative CRC treatment (postoperatively and post adjuvant chemotherapy) to identify the best-performing method at each time point.

S2: To assess the effect of standard-of-care adjuvant chemotherapy on the level of ctDNA. Especially, for patients with ctDNA detected after surgery, the aim is to measure and compare the ctDNA levels in plasma samples drawn before and after adjuvant chemotherapy. Further, the change in ctDNA level will be correlated to the oncological outcomes (time to clinical recurrence, disease-free survival, and overall survival).

S3: To investigate if time to Molecular recurrence determined using serial ctDNA analyses in longitudinally collected plasma samples is shorter than time to Clinical recurrence using standard-of-care radiological imaging.

S4: To investigate the correlation between ctDNA analysis results and findings on CT scans. ctDNA analysis will be restricted to blood sampling times that coincide with standard-of-care CT scans (at 12 and 36 months postoperatively). If ctDNA analysis can predict the outcome of the CT scan, the potential is that ctDNA analysis in the future can guide when to perform CT scans.

S5: To investigate the prognostic power of ctDNA at the time point of indeterminate CT scans.

S6: To investigate, if molecular characterization of CRC cancers can stratify patients and predict i.e., treatment response, growth patterns, cancer aggressiveness, clinical outcomes, and whether the tumor sheds ctDNA into the circulation.

Investigational plan

The DANISH.MRD study is logistically divided into two parts, and patients are offered participation in each part separately. The parts are called "DANISH.MRD part I - Surgery", and "DANISH.MRD part II - Surveillance".

In DANISH.MRD part I blood samples are collected before and after surgery. For patients receiving neoadjuvant therapy, a blood sample will also be collected before initiation of this treatment.

In DANISH.MRD part II blood samples are collected immediately after adjuvant chemotherapy and during standard-of-care surveillance.

Patients included in DANISH.MRD part I will help address Primary objective 1 (P1). The subset of the part I patients that are also included in DANISH.MRD part II will help to address the Secondary objectives S1-S6.

Both Part I and Part II DANISH.MRD patients receive standard follow-up care, which includes scheduled visits for up to 5 years following their surgery.

Sample collection for DANISH.MRD part I - Surgery (Objectives P1-2, S1-S5)

* Blood sampling preoperatively and after surgery (between days 20-30, but before initiation of adjuvant chemotherapy)
* Sampling of tissue from the resected specimen

Sample collection in DANISH.MRD part II - Surveillance (objectives S1-S5)

* Blood sampling post-adjuvant chemotherapy (ACT): postACT (14-30 days after the end of ACT), and at months 8, 12, 16, 20, 24, 30 and 36 postoperatively.

ELIGIBILITY:
DANISH.MRD part I - Surgery

Inclusion Criteria:

* Colon or rectal cancer, clinical tumor stage I-III.
* Patient able to understand and sign written informed consent.
* Scheduled for curative-intent resectional surgery (including "compromised" curative resections).

Exclusion Criteria:

* Hereditary colorectal cancer linked to familial colonic polyposis or Lynch syndrome.
* Inflammatory bowel disease (Crohn's disease or ulcerative colitis).
* Verified distant metastases.
* Malignant colorectal polyps diagnosed after polypectomy.
* Patients who are unlikely to comply with the protocol (e.g., uncooperative attitude, inability to return for subsequent visits) and/or otherwise considered by the Investigator to be unlikely to complete the study.

DANISH.MRD part II - Surveillance

Inclusion Criteria:

* Participation in DANISH.MRD part I - Surgery.
* Colorectal cancer, UICC stage III.
* Has received curative-intent resection and is a candidate for adjuvant chemotherapy (3- or 6-months regime).

Exclusion Criteria:

* Not treated with adjuvant chemotherapy
* Treated with neoadjuvant chemo-radiation therapy.
* Synchronous colorectal and non-colorectal cancer diagnosed per operative (except skin cancer other than melanoma).
* Other cancers (excluding colorectal cancer or skin cancer other than melanoma) within 3 years from eligibility screening.
* Patients who are unlikely to comply with the protocol (e.g., uncooperative attitude, inability to return for subsequent visits) and/or otherwise considered by the Investigator to be unlikely to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: DANISH.MRD part I - Surgery Patients with colorectal cancer clinical stage I-III scheduled for curative-intent resectional surgery.
  DANISH.MRD part I - Surveillance Patients participating in DANISH.MRD part 1, and pathological stage III colorectal cancer, and candidates for adjuvant chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2028-07-30 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
The prognostic value of ctDNA status | 3 years after surgery
  Especially, the association between 3-year disease-free survival and ctDNA status after surgery and after adjuvant chemotherapy

SECONDARY OUTCOMES:
Ranking of commercial ctDNA diagnostics | 3 years after surgery
  Technical assessment to compare and rank commercial ctDNA diagnostics and evaluate their performance after surgery and adjuvant chemotherapy
Change in ctDNA levels after adjuvant chemotherapy | 3 years after surgery
  Assessment of the effect of standard-of-care chemotherapy on the level of ctDNA
Lead time between molecular and clinical recurrence | 3 years after surgery
  Assessment of the time between molecular recurrence (ctDNA positive blood sample) and clinical recurrence (standard-of-care radiological imaging)
Correlation between ctDNA analysis and findings on CT scans | 3 years after surgery
  ctDNA status on blood samples coinciding with standard-of-care CT scans (at 1 and 3 years after surgery), to see if ctDNA analysis can predict the outcome of the CT scan
Prognostic power of ctDNA at the time point of an indeterminate CT scan | 3 years after surgery
Molecular characterization | 3 years after surgery
  Investigation of the use of molecular characterization to stratify patients and predict i.e., treatment response, growth patterns, cancer aggressiveness, clinical outcomes, and whether the tumor sheds ctDNA into the circulation

CONTACTS AND LOCATIONS:
Overall Officials: Claus L Andersen, PhD, Principal Investigator — Aarhus University Hospital; Lene H Iversen, MD, DMSc, Principal Investigator — Aarhus University Hospital; Kåre A Gotschalck, MD, PhD, Principal Investigator — Regionshospitalet Horsens
Locations (10):
- Denmark (10):
  - Bispebjerg Hospital, Copenhagen, Capital Region of Denmark
  - Herlev Hospital, Herlev, Capital Region of Denmark
  - Aarhus University Hospital, Aarhus, Central Jutland
  - Gødstrup Hospital, Herning, Central Jutland
  - Regional Hospital Horsens, Horsens, Central Jutland
  - Regional Hospital Randers, Randers, Central Jutland
  - Regional Hospital Viborg, Viborg, Central Jutland
  - Aalborg University Hospital, Aalborg, North Denmark
  - Odense University Hospital, Odense, The Region of Southern Denmark
  - Vejle Hospital, Vejle

IPD SHARING:
Plan to Share IPD: No